CLINICAL TRIAL: NCT04446078
Title: Hybrid Polyetheretherketone (PEEK)-Acrylic Resin Prostheses and the All-on-4 Concept for Full Arch Rehabilitation
Acronym: AO4PEEKDev
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Malo Clinic (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: AO4PEEKDevGroup
Record Dates: First submitted 2020-06-22; First posted 2020-06-24 (Actual); Last update posted 2023-02-24 (Actual); Status verified 2023-02

CONDITIONS: Dental Implants; Dental Materials; Mandible; Prosthesis Survival
Keywords: All-on-4; All-on-four
MeSH Terms: conditions — Prosthesis Failure

STUDY DESIGN:
Intervention Model Description: prospective cohort
Masking Description: patient coding
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- PEEK - All-on-4 (Experimental): Patients rehabilitated with a PEEK-acrylic resin prosthesis supported by immediate function dental implants inserted through the All-on-4 concept
  Interventions: Device: PEEK- acrylic resin prosthesis supported by 4 dental implants

INTERVENTIONS:
Device: PEEK- acrylic resin prosthesis supported by 4 dental implants — Patients rehabilitated for edentulism of one or both arches through an implant supported fixed prosthesis

SUMMARY:
It is necessary to evaluate the outcome of implant supported fixed prosthetic rehabilitations using peek material. To test this, the study design to be used will be a prospective single cohort to evaluate the long term outcome of fixed prosthetic implant supported rehabilitations. The cohort will be evaluated after 5 years of follow-up, regarding prosthetic survival, implant survival, marginal bone resorption, incidence of mechanical complications (loosening or fracture of prosthetic components), biological complications (peri-implant pathology, suppuration, fistulae), incidence of biological complications (peri-implant pathology, suppuration, excessive marginal bone resorption) in-mouth comfort, overall chewing feeling, framework integrity, veneer adhesion, veneer chipping, patient tissue reaction, denture staining, manufacture issues,

DETAILED DESCRIPTION:
Problem Peek material is already used in the dentistry field, but proof on its long-term outcome in implant supported fixed rehabilitations is lacking.

Objectives

* To evaluate the long term outcome of fixed prosthetic implant supported rehabilitations using peek material.
* To report the results.

Significance This investigation is of interest, because it will provide an overview of the long term outcome of implant supported fixed prosthetic rehabilitations using peek material.

Hypothesis The hypothesis that this study will evaluate, will be the distribution of survival and other variables of interest in implant supported fixed prosthetic rehabilitations using peek material.

Materials and Methods Methodology This study will be performed at Malo Clinic in Lisbon. It is estimated to last for approximately 5 years. The study design to be used will be a prospective single cohort study to evaluate the long-term outcome of implant supported fixed prosthetic rehabilitations using peek material. The cohort will be evaluated in at least 5 interventions (1 per year), regarding survival and the clinical/technical parameters established in this study. There will be no risk for the participants, has all procedures for collecting information will be minimally invasive and non- traumatizing.

Population The population of this study consists in individuals rehabilitated with a fixed prosthetic rehabilitation supported by immediate function implants, of both genders, without age restrictions.

Sample size It is expected that the sample will consist of 37 consecutively treated patients during the year of 2013.

External variables:

* Withdrawal of the patients;
* The patient missing the control appointment;
* Interruption of the treatment by the patient;
* Patient deceased.

Statistical analysis:

In this study, the data will be treated by means of descriptive and inferential statistics. The data will be treated using the Statistical Package for Social Sciences (SPSS) for Windows version 17.0 ®. Survival will be estimated through life tables. Inferential analysis will be performed for characterization of the cohort and independent variables.

Adverse events:

An adverse event is defined as any undesirable clinical occurrence in a subject whether it is considered to be device related or not. If the adverse event is regarded as device related it is stated as an adverse device effect. An adverse event or adverse device effect may be serious\severe or non-serious\non-severe. If, as result of an adverse event during a clinical investigation, a subject has to be hospitalized, or their hospitalization is unduly prolonged due to potential disability or danger to life because an intervention has been necessitated or the event is terminal, the adverse event or adverse effect is regarded as serious. All serious adverse events must be reported to the Ethic Committee and without any delay.

Ethical aspects:

This investigation will be carried out in accordance to the ethical principles and guidelines stated in the Declaration of Helsinki. The Investigation should be evaluated and approved by a National Ethic Committee prior to including the first subject in the investigation. The application to the Ethic committee is to be made by the responsible investigators, and a copy of the approval should be sent to the monitor before the investigation starts. It is also of great importance that each subject receives oral and written information about the investigation, and that she/he must only participate if they truly want to do so. Also, the subjects must be aware of the fact that they can withdraw from the investigation at any time and for any reason without jeopardizing their future treatment.

Furthermore, the subjects should be made aware of the fact that the data from his/her treatment will be registered in a computer database, but that she/he will only be registered through a code system. This means that the identity of each subject will be unknown to all others than the doctor performing the treatment. Each subject is entitled to take part of the information stored about her/his treatment. This information is to be handed out by the treating doctor.

Database management:

The data collected from the forms will be introduced in a digital database (Microsoft Office Excel 2003®). The database management will be the responsibility of the Malo Clinic.

ELIGIBILITY:
Inclusion Criteria:

* rehabilitated with implant-supported fixed prostheses through the All-on-4 concept (Nobel Biocare)

Exclusion Criteria:

* Patients in active chemotherapy or radiotherapy,
* Presenting insufficient bone volume,
* Unable to provide written informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 37 (Actual)
Dates: Start 2014-05-02 (Actual); Primary Completion 2021-12-29 (Actual); Study Completion 2022-02-09 (Actual)

PRIMARY OUTCOMES:
prosthetic survival | 5 years
  considering the necessity of replacing the prosthesis; fracture of the infrastructure

SECONDARY OUTCOMES:
implant survival | 5 years
  considering the implants' function, censoring as a failure the first implant to fail in a given patient
marginal bone loss | 5 years
  Marginal bone level was defined as the distance between the implant's platform and the most apical bone-implant contact, while the measurements difference between baseline (connection of the definitive prosthesis) and the subsequent evaluation.
Plaque levels | 5 years
  modified plaque index
Bleeding levels | 5 years
  modified bleeding index
Problems during manufacturing | 5 years
  Evaluation of veneer adhesion by detachment of acrylic resin veneer from PEEK infrastructure.
Biological complications | 5 years
  Adverse soft tissue reaction, suppuration, abscess, fistulae and peri-implant pathology (the presence of marginal bone loss and peri-implant pockets of more than 4 mm, with or without the concurrent presence of bleeding on probing or suppuration)
Mechanical complications | 5 years
  Prosthesis, abutments or prosthetic screws fracture or loosening
Patient subjective evaluation concerning overall chewing feeling associated with the specific feel during food mastication | 5 years
  The evaluations performed by the patient were registered on a visual analogue scale ranging between 0-10 (poor to excellent)
Patient subjective evaluation concerning in mouth comfort specified as the patients' overall evaluation according to the expectations when submitting the prosthesis to function | 5 years
  The evaluations performed by the patient were registered on a visual analogue scale ranging between 0-10 (poor to excellent)

CONTACTS AND LOCATIONS:
Overall Officials: Miguel A de Araújo Nobre, PhD, Principal Investigator — Malo Clinic
Locations (1):
- Malo Clinic, Lisbon, Portugal

IPD SHARING:
Plan to Share IPD: No